CLINICAL TRIAL: NCT00443742
Title: Diagnosis of Depression Among Adolescents - a Clinical Validation Study of Key Questions and Questionnaire
Brief Title: Diagnosis of Depression Among Adolescents
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Other Study IDs: S-06293a
Record Dates: First submitted 2007-03-03; First posted 2007-03-06 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Depression
Keywords: Depression; Validation; Adolescent; Validation of three key questions and questionnaire
MeSH Terms: conditions — Depression | interventions — Validation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Validation

SUMMARY:
The objective of the study is to improve general practitioners' diagnoses of adolescent depression. Major depression is ranked fourth in the worldwide disability impact. The proportion of adolescents suffering from depressive disorders also seems to be increasing worldwide. Early interventions are known to reduce this illness. Therefore, the earlier depression can be identified in adolescents, the greater the advantage.

ELIGIBILITY:
Inclusion Criteria:

* age (14-16)

Exclusion Criteria:

* not fluency in the Norwegian and Danish language

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 323 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Rikard Haavet, MD, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway